CLINICAL TRIAL: NCT05145569
Title: A Phase 2 Open-label Study to Assess the Antitumor Activity of Neoadjuvant Chemotherapy with or Without HCW9218 in Patients with Metastatic Advanced Stage Ovarian Cancer
Brief Title: Antitumor Activity of Neoadjuvant Chemotherapy with or Without HCW9218 in Metastatic Advanced Stage Ovarian Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Per PI and agent sponsor
Sponsor: Haider Mahdi (Other)
Collaborators: HCW Biologics (Industry)
Responsible Party: Sponsor-Investigator, Haider Mahdi, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 21-162
Record Dates: First submitted 2021-11-22; First posted 2021-12-06 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Ovarian Cancer
Keywords: TGFβ receptor II (TGFβRII or TGFβ Trap); PD-L1
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carboplatin/paclitaxel + HCW9218 (Experimental): HCW9218 in combination with chemotherapy including carboplatin AUC 5 and paclitaxel 175 mg/m2 on Day 1 of the 21-day cycle
  Interventions: Drug: Carboplatin AUC 5 and paclitaxel; Drug: HCW9218
- Carboplatin/paclitaxel (Active Comparator): Carboplatin AUC 5 and paclitaxel 175 mg/m2 on Day 1 of the 21-day cycle
  Interventions: Drug: Carboplatin AUC 5 and paclitaxel

INTERVENTIONS:
Drug: Carboplatin AUC 5 and paclitaxel — Carboplatin AUC 5 and paclitaxel combination chemotherapy is very well tolerated and highly effective for the treatment of ovarian cancer and thus is standard of care therapy. Both carboplatin and paclitaxel are chemotherapy agents that are designed to kill and slow the growth of cancer cells.
  Other Names: Carbo/Taxol
Drug: HCW9218 — HCW9218 is an immunotherapeutic comprising transforming growth factor-b (TGF-b) receptor II and interleukin (IL)-15/IL-15 receptor a domains.
  Arms: Carboplatin/paclitaxel + HCW9218

SUMMARY:
In this study, the safety, tolerability, and anti-tumor activity of HCW9218 in combination with chemotherapy will be assessed in patients with advanced stage ovarian cancer undergoing neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Existing data supports a potential role and synergistic activity between TGF-β inhibitors and PD1 TGF-β has been investigated in ovarian cancer and it is suggested to play a dominant role as a potent inducer of ovarian cancer invasiveness and metastasis in additional studies [36]. In fact, TGF-β ligand and TGF-β receptor I and II are strongly expressed in ovarian tumors especially high-grade ovarian cancers. Further, TGF-β is abundantly secreted into the tumor microenvironment by cancer and stromal cells in this cancer. TGF-β expression has been shown to significantly higher in ovarian cancer tissue especially advanced stage disease compared to healthy tissue or borderline tumors. Inhibiting senescence in the immune compartment may have a profound effect on the cytotoxic functions of both innate and adaptive immune cells. This study aims to examine markers of senescence on immune cells obtained from blood throughout the proposed trial. We hypothesize that HCW9218 will act as a senolytic by "trapping" excess TGF-β, therefore inhibiting its ability to promote senescence. We believe that this combined with the immune activating effect of IL-15 will be a biologically relevant therapeutic with potential to at least partially reverse therapy induced senescence (TIS) or in the future, perhaps have an effect even on physiologic aging.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of ovarian cancer who meets below inclusion criteria will be enrolled in this study.
2. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
3. Provision of signed and dated, written informed consent form prior to any mandatory study specific procedures, sampling, and analyses.
4. A female participant is eligible to participate if she is not pregnant (see Appendix E), not breastfeeding, and at least one of the following conditions applies:

d1. Not a woman of childbearing potential (WOCBP) as defined in Appendix E

d2. A WOCBP who agrees to follow the contraceptive guidance in Appendix E during the treatment period and for at least 120 days after the last dose of study treatment.

Diagnosis/Condition for Entry into the Trial:

1. World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1 or 2 at enrollment.
2. Must have a life expectancy of at least 12 weeks
3. Patients with histologically or cytologically confirmed epithelial ovarian, fallopian or primary peritoneal cancer. patients should have diagnosis of advanced stage (III-IV) ovarian cancer who are planned to have neoadjuvant chemotherapy with carboplatin and paclitaxel.
4. High grade serous histology
5. Patients have to be chemo-naïve with no prior chemotherapy or any therapy for ovarian cancer.
6. Confirmation of measurable disease based on RECIST 1.1 by investigators at Screening will be used to determine patient eligibility and imaging shows at least 1 lesion that is appropriate for selection as a target lesion per RECIST 1.1 is required prior to patient treatment. Tumor assessment by computed tomography (CT) scan or magnetic resonance imaging (MRI) must be performed within 28 days prior to C1D1.
7. All patients enrolled must be ICI-naïve patients defined as no prior exposure to immune-mediated therapy including, but not limited to, other anti CTLA-4, anti-PD-1, anti-PD-L1, and anti-programmed cell death ligand 2 (anti-PD-L2) antibodies, excluding therapeutic anticancer vaccines.
8. All patients must be able to provide a tumor tissue either archival tissue or newly acquired tumor biopsy. The tumor specimen should be of sufficient quantity to allow for exploratory biomarker analyses.
9. Have adequate organ function as defined in Table 1. Specimens must be collected within 7 days prior to the start of study treatment.

Exclusion Criteria:

Pregnancy Exclusion:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation (see section 6.4 Pregnancy Testing). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
3. Is pregnant or breastfeeding or expecting to conceive within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.

Prior/Concurrent Clinical Study Experience:

1. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

Note: Patients who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

Prior/Concomitant Therapy:

1. Has received prior therapy with a TGF-β antagonist, IL-15 or analogs.
2. Has received prior systemic anti-cancer therapy including investigational agents prior to treatment. Note: Patients must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Patients with ≤Grade 2 neuropathy may be eligible. Note: If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
3. Has received prior radiotherapy within 2 weeks of start of study treatment. Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
4. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
5. Known severe hypersensitivity (Grade ≥ 3 NCI CTCAE 5.0) to compounds of similar chemical or biologic composition to the investigational product used in the study or any component in its formulations, any history of anaphylaxis, or recent, within 5 months, history of uncontrollable asthma.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.

Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

Medical conditions:

1. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
2. Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.

   Note: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in-situ cancers
3. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
4. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
5. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
6. Has an active infection requiring systemic intravenous therapy.
7. Has a known history of human immunodeficiency virus (HIV) infection or HIV test (+) in screening test. No HIV testing is required unless mandated by local health authority. Patients with HIV infection with following exception are allowed: HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of enrollment are eligible for this trial.
8. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection except following situation: Patients with a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection are allowed to be included if: participant on a stable dose of antiviral therapy, HBV viral load below the limit of quantification. HCV viral load below the limit of quantification.
9. Has a known history of active tuberculosis (TB).
10. History of bleeding diathesis or recent major bleeding events (i.e., Grade ≥ 2 bleeding event the month prior treatment).
11. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III/IV), uncontrolled hypertension (≥150/90mmHg), unstable angina pectoris or myocardial infarction (≤ 6 months prior to screening), uncontrolled cardiac arrhythmia, clinically significant cardiac valvulopathy requiting treatment, active interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
12. QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥450 ms in male and ≥470 ms in female calculated from 12-lead ECGs.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety - Dose Limiting Toxicities (DLT) | Up to 8 weeks
  A Dose Limiting Toxicity (DLT) is defined hematologic or non-hematologic toxicity (assessed in accordance with NCI CTCAE v 5.0), clearly attributable to HCW9218 (experimental agent) which cause any immune-related grade 3 or grade 4, or recurrent grade 2 toxicities, requiring discontinuation of HCW9218 or treatment delay for more than 4 weeks.
  The criteria for stopping will be P(P(DLT)>0.2)>0.66, which will be evaluated after every 5 patients on the chemotherapy plus HCW9218 arm have completed their safety observation period (four cycles). The probability statement will be assessed using a beta-binomial rule with a prior that assumes unacceptable toxicity will occur in 10% of patients (α=1 and β=9).
Adverse Events Related to Treatment | Up to 12 months
  Incidence, nature and severity of adverse events (AEs) graded according to NCI CTCAE v5.0.
Complete Pathologic Response | Up to 36 months
  Proportion of patients that experience a complete absence of cancer after study treatment as determined by pathological/histological assessment of tissue samples.
CD8+ T-cell characterization | Up to 12 months
  CD8+ T-cell infiltration and other alterations in tumor immune microenvironment.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) at 6 months | Up to 6 months
  The proportion of patients who remain progression-free from the initial date of treatment until 6 months afterwards, with progression defined by RECIST v1.1.Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Progression-free Survival (PFS) at 12 months | Up to 12 months
  The proportion of patients who remain progression-free from the initial date of treatment until 12 months afterwards, with progression defined by RECIST v1.1.Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Progression-free Survival (PFS) at 18 months | Up to 18 months
  The proportion of patients who remain progression-free from the initial date of treatment until 18 months afterwards, with progression defined by RECIST v1.1.Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Progression-free Survival (PFS) | Up to 5 years
  Progression-free survival is the median (estimated) time measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression),whichever occurs first, with progression defined by RECIST v 1.1.Progressive disease(PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Overall Survival (OS) at 6 months | Up to 6 months
  The proportion of patients that remain alive from the start of treatment until death from any cause at 6 months.
Overall Survival (OS) at 12 months | Up to 12 months
  The proportion of patients that remain alive from the start of treatment until death from any cause at 12 months.
Overall Survival (OS) at 18 months | Up to 18 months
  The proportion of patients that remain alive from the start of treatment until death from any cause at 18 months.
Overall Survival (OS) | Up to 5 years
  The median length of time (estimated) from the start of treatment that patients remain alive, until death from any cause.
Duration of Response (DOR) | Up to 36 months
  Time from first confirmation of response to evidence of disease progression. Progression defined by RECIST v 1.1.Progressive disease(PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time to Tumor Response (TTR) | Up to 36 months
  Time from trial enrollment to first documentation of objective response per RECIST v1.1. Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Disease Control Rate (DCR) | Up to 36 months
  The proportion of treated with Complete Response (CR) + Partial Response (PR) + Stable Disease (SD), per RECIST v1.1. Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. Stable Disease (SD) is defined as neither sufficient shrinkage (compared to baseline) to qualify for partial or complete response (CR or PR) nor sufficient increase (taking as reference the smallest sum of diameters at baseline or while on study, whichever is smallest) to qualify for progressive disease (PD).
Objective Response Rate (ORR) | Up to 36 months
  The proportion of treated patients with Complete Response (CR) + Partial Response (PR), per RECIST v1.1. Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Stable Disease at 12 weeks | At 12 weeks
  Per RECIST v1.1, Stable Disease (SD) is defined as neither sufficient shrinkage (compared to baseline) to qualify for partial or complete response (CR or PR) nor sufficient increase (taking as reference the smallest sum of diameters at baseline or while on study, whichever is smallest) to qualify for progressive disease (PD).

CONTACTS AND LOCATIONS:
Overall Officials: Haider S Mahdi, MD, Principal Investigator — UPMC Hillman Cancer Center

IPD SHARING:
Plan to Share IPD: No